CLINICAL TRIAL: NCT07296588
Title: Expert Consensus on Photoprotection Practices: A Delphi Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Venus Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: Photoprotection-VRC
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Photoprotection; Sunscreen; Sunscreen Agents; Sun Damaged Skin; Sun Exposure
Keywords: Photopretection; sunscreen; consensus; delphi method; Expert panel

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert Panel: The study population will consist of a purposive sample of dermatologists, photobiologists, and other experts actively involved in photoprotection research, clinical practice, or public health initiatives. Panelists should have experience advising patients or the public on sunscreen use, UV protection strategies, or photodermatoses.
  Panel Size and Rationale:
  Target enrollment: 20-35 experts
  Large enough to capture diverse perspectives while remaining feasible for iterative Delphi rounds.
  Minimum for analysis: 15 panelists to ensure adequate representativeness in case of attrition.

SUMMARY:
This study is a Delphi-based expert consensus project aimed at developing evidence-informed recommendations for photoprotection practices across various populations, including general, at-risk, and special groups (e.g., children, pregnant women, patients with photodermatoses). Despite extensive evidence on the importance of sun protection, there is variability in clinical advice regarding sunscreen selection, application frequency, SPF requirements, adjunctive protective measures, and patient counseling.

DETAILED DESCRIPTION:
This study is a non-interventional, methodological Delphi consensus project designed to develop standardized recommendations for photoprotection practices. Photoprotection encompasses strategies to minimize ultraviolet (UV)-related skin damage, including sunscreen use, clothing, behavioral measures, and patient education. Despite broad awareness campaigns, inconsistencies exist regarding SPF selection, application methods, timing, reapplication frequency, and the use of additional protective measures.

A steering committee of dermatologists and photoprotection experts will conduct a literature review and draft initial statements addressing key domains:

Sunscreen use: SPF level, spectrum coverage (UVA/UVB), formulation (chemical vs. physical), water resistance.

Application guidelines: Amount, timing before sun exposure, reapplication frequency, body coverage.

Adjunctive measures: Protective clothing, hats, sunglasses, shade-seeking behavior.

Special populations: Children, pregnant women, outdoor workers, patients with photosensitive dermatoses.

Behavioral counseling: Education strategies, adherence promotion, and misconceptions.

Integration with skin care and aesthetic practices.

A panel of experts in dermatology, photobiology, and related fields will participate in multiple Delphi rounds. Panelists will rate agreement with each statement using a Likert scale. Anonymized feedback will be provided after each round, and statements not reaching a predefined consensus threshold (e.g., ≥70-80%) will be revised and re-evaluated in subsequent rounds.

The final output will consist of consensus-based recommendations reflecting practical, safe, and evidence-informed photoprotection practices. Areas of disagreement or uncertainty will also be highlighted, identifying research gaps and priorities for future studies.

ELIGIBILITY:
Inclusion Criteria:

Board-certified dermatologists, photobiologists, or clinicians/researchers with ≥5 years of relevant experience.

Regular involvement in advising on photoprotection, skin cancer prevention, or UV-related dermatology.

Engagement in research, guideline development, teaching, or professional society activities related to dermatology, photobiology, or public health.

Willingness and availability to participate in all Delphi rounds.

Exclusion Criteria:

* Non-dermatology or non-photobiology specialists without relevant experience.

Less than 5 years of relevant clinical or research experience.

Limited or no experience with photoprotection counseling or research.

Significant undisclosed conflict of interest related to sunscreen or photoprotection products.

Inability or unwillingness to participate in all Delphi rounds.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of a purposive sample of experts in dermatology, photobiology, and related fields who are actively involved in photoprotection research, clinical practice, or public health initiatives. Panelists should have experience advising patients or populations on sun protection, sunscreen use, and UV-related skin care.
  Panel Size and Rationale:
  Target enrollment: 20-35 experts
  Sufficient to capture diverse perspectives while remaining manageable for multiple Delphi rounds.
  Minimum for analysis: 15 panelists, ensuring representativeness in case of attrition
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 6-12 weeks
  Level of expert consensus on statements regarding photoprotection practices, measured as the proportion of panelists reaching the predefined agreement threshold (e.g., ≥70-80%) per statement across Delphi rounds.

SECONDARY OUTCOMES:
Secondary Outcomes | 6-12 weeks
  Consensus on sunscreen use: SPF level, broad-spectrum coverage, formulation, and water resistance.
  Consensus on application guidelines: amount, timing before sun exposure, reapplication frequency, body coverage.
  Consensus on adjunctive measures: protective clothing, hats, sunglasses, shade-seeking behavior.
  Consensus on special populations: children, pregnant women, outdoor workers, photosensitive patients.
  Consensus on behavioral counseling and education strategies for adherence.
  Identification of areas of uncertainty requiring further research or regional adaptation.

CONTACTS AND LOCATIONS:
Locations (1):
- Venus Research Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Delphi studies do not collect patient data, medical records, biological samples, or identifiable clinical information. Experts only give opinions, not "IPD." Their responses are anonymized, and sharing identifiable expert-level responses is not required and often discouraged